CLINICAL TRIAL: NCT01121081
Title: A Randomized, Double-Blind, , Placebo Controlled, 18 Week Study To Evaluate the Efficacy of Adjuvant 9-cis-β-Carotene Rich Powder of the Alga Dunaliella Bardawil in Subjects With Plaque Type Psoriasis Treated by Narrow Band UVB Therapy
Brief Title: The Effect of Algae Dunaliella Bardawil on Psoriasis (2)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: no patients enrolled
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: The Bert W. Strassburger Lipid Center, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHEBA-09-7464-FP-CTIL
Record Dates: First submitted 2010-04-11; First posted 2010-05-12 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Psoriasis
Keywords: Male or female subjects; ≥18 to ≤75 years of age; who have a diagnosis of plaque or guttate psoriasis
MeSH Terms: conditions — Psoriasis; Guttate Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): sugar pills
  Interventions: Drug: Placebo
- Dunaliella (Experimental): drug
  Interventions: Drug: Alga Dunaliella Bardawil

INTERVENTIONS:
Drug: Alga Dunaliella Bardawil — 4 capsules per day, 2 in the morning 2 in the evening for 3 month
  Other Names: Active Comparator
  Arms: Dunaliella
Drug: Placebo — Drug: Alga Dunaliella Bardawil
  4 capsules per day, 2 in the morning 2 in the evening for 3 month
  Other Names: Placebo Comparator
  Arms: Placebo

SUMMARY:
This is a Randomized, Double-Blind, , Placebo Controlled, 18 Week Study To Evaluate the Efficacy of adjuvant 9-cis-β-Carotene Rich powder of the Alga Dunaliella bardawil in Subjects With Plaque type Psoriasis treated by Narrow Band UVB therapy.

DETAILED DESCRIPTION:
This is a double blind, parallel group, randomized study with 12 weeks of daily oral administration of Dunaliella or placebo in psoriasis patients undergoing phototherapy.

Subjects will be screened for eligibility at the baseline visit for phototherapy and blood tests.

After screen phase of maximum two weeks the subjects will be randomized at phototherapy treatment no. 4 in to one of two treatments groups (2:1): Dunaliella or placebo.

Each subject will have a final evaluation 4 weeks after the end of study drug treatment .

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet ALL of the following criteria will be considered for enrollment into this study:

  1. Signed and dated written Institutional Review Board (IRB) or Independent Ethics Committee (IEC) approved informed consent obtained from the subject in accordance with the local regulations;
  2. Male or female subjects, ≥18 to ≤75 years of age, who have a diagnosis of plaque or guttate psoriasis;
  3. Psoriasis Area and Severity Index (PASI) score of ≥12 or psoriasis covering ≥10% of body surface area (BSA)
  4. Psoriasis severity at least moderate, scoring at least 3 on the 0 to 5 point Physician Global Assessment (PGA) scale of the National Psoriasis Foundation Psoriasis Score (NPF-PS)
  5. Candidate to phototherapy treatment starting at visit 0.
  6. For a female subject; either:
* subject is non-childbearing potential, defined as: menopause with amenorrhea >2 years, hysterectomy, or bilateral oophorectomy or
* agrees to continue to use adequate contraception (i.e., hormonal [oral, depot, patch], IUD, barrier and spermicide) throughout the study and for at least one month following termination and have a negative urinary pregnancy test at screening and before the first dose of study drug; 7. In the opinion of the investigator, the subject will be compliant and have a high probability of completing the study and all required procedures.

Exclusion Criteria:Subjects who meet ANY of the following criteria will be excluded from participation in this study:

1. The subject presents with the predominant type of psoriasis as erythrodermic, inverse, pustular or pulmo-plantar or an unstable form of psoriasis;
2. Received any investigational drug within 30 days of randomization.
3. The subject has not undergone wash-out periods of sufficient duration for the following treatments at Baseline:

   Topical psoriasis treatments: 2 weeks Systemic psoriasis treatments: 4 weeks or 5 half lives (whichever is longer) Phototherapy or climatotherapy : 4 weeks Biologic treatments: 4 weeks
4. The subject anticipates getting enough extra trial ultra-violet light during the study (e.g. sunbathing; tanning salon, etc.) to cause psoriasis to improve;
5. The subject has a known allergy or sensitivity to the study treatment(s) or to any of the participant contained in the study drug formulation
6. Any other acute or chronic medical condition that, in the opinion of the investigator, increases the risk to the subject or the likelihood that the subject will be unable to complete the study;
7. Subjects with any laboratory test at screening considered significantly abnormal.

   The following will be considered significantly abnormal:

   Alanine transaminase (ALT), aspartate transaminase (AST) > 3 upper limit normal. CPK > 3 upper limit normal. Triglycerides > 350mg/dl.

   cytopenia (to include any of the following: WBC <3.5x10 3/μL; Hgb <10 g/dL; platelets <120x10 3/μL; neutrophils absolute <1.5x10 3/μL; lymphocytes absolute <0.8x10 3/μL) or
8. Personal or first degree relative history of malignant melanoma.
9. Known serologic positivity for human immunodeficiency virus or hepatitis B or C virus.
10. History of substance abuse, including alcohol abuse, within the past year.
11. History or current clinically significant major psychiatric disorder (e.g., major depressive disorder, psychosis, schizophrenia) according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM IV TR) [Exception; subjects with depression that has been adequately controlled for at least 6 months may enroll in the study];
12. Female subject with a positive pregnancy test or nursing, or planning a pregnancy during the course of the study;
13. Unwilling or unable to comply with study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index (PASI)75% | 3 month
  Patient disease and skin condition will be assessed using Psoriasis Area and Severity Index and compared to condition on baseline, The PASI score will be calculated at each visit

SECONDARY OUTCOMES:
PASI 50 | 3 month
  The PASI 50 is an assessment of the proportion of patients who achieve at least 50% improvement in the PASI score from baseline Psoriasis Area and Severity Index (PASI)will be calculated at each visit
Durability of Response | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Felix Pavlotsky,, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel